CLINICAL TRIAL: NCT06420921
Title: MeasurIng and Restoring Auditory Awareness for Cochlear Implant Listeners in noisE
Acronym: MIRACLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de l'Audition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-153
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Noise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with cochlear implant (Experimental)
  Interventions: Behavioral: Speech in noise comprehension test; Behavioral: Objective tests of perception of ambient sound cues in noise; Behavioral: Subjective tests of perception of ambient sound cues in noise
- Normal hearing participants (Active Comparator)
  Interventions: Behavioral: Speech in noise comprehension test; Behavioral: Objective tests of perception of ambient sound cues in noise; Behavioral: Subjective tests of perception of ambient sound cues in noise

INTERVENTIONS:
Behavioral: Speech in noise comprehension test — Speech in noise comprehension tests consisting of listening to a speech source and one or more competing sources (noise, speech or sound cues) simultaneously. The volunteers will have to repeat the speech source in order to assess intelligibility for each situation, as a function of the intensity ratio of the two sources (SNR).
Behavioral: Objective tests of perception of ambient sound cues in noise — Tests of perception of the sound environment consisting of listening to a source of noise, sound cues and a competing source of speech simultaneously. The volunteers will have to identify sound cues in order to assess the ability to perceive the sound environment for each situation, depending on the intensity ratio of the different sources.
Behavioral: Subjective tests of perception of ambient sound cues in noise — Tests of perception of the sound environment consisting of listening to a source of noise, sound cues and a competing source of speech simultaneously. Using a simple interface, the volunteers will have to identify the intensity ratio of the sources that they consider to be the best compromise between understanding speech and perceiving the sound environment.

SUMMARY:
The goal of this interventional study is to describe how people with cochlear implants perceive the perceive speech in noise and their sound environment on adults who are native French speakers with typical hearing or with cochlear implant(s).

The measures and strategies developed in this project could benefit all current and future cochlear implant wearers by improving their perception of the sound environment and their quality of life on a daily basis.

Researchers will compare normal hearing participant and participants with cochlear implant to describe the speech in noise and their perception of the sound environment.

Participants will perform audiological tests to assess their perception of the sound environment, with and without speech enhancement.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* 18 years of age or over,
* Native French speaker,
* Having given their consent to take part in the research.

For cochlear implant patients:

* Adult implanted and declaring that they have been using the implant for at least 18 months,
* Normal speech audiometry in silence

For controls reporting normal hearing:

* Normal tonal audiometry (defined as a mean tonal loss not exceeding 30 decibel (dB) HL)
* Normal speech audiometry in noise (SNR between -8 dB and -4dB inclusive)

Exclusion Criteria:

* Be under guardianship or curatorship,
* deprived of liberty by judicial or administrative decision, or subject to legal protection,
* Non- native French speaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
percentage of environmental sound cues correctly identified when presented simultaneously with other signals | 2 years

SECONDARY OUTCOMES:
comparison of the percentages of correctly identified environmental sound cues obtained objectively and deduced from the signal-to-noise ratio corresponding to the trade-off indicated by the participant | 2 years
the percentages of words correctly repeated by participants using non-personalised speech enhancement strategies | 2 years
percentages of words correctly repeated by participants using personalised speech enhancement strategies | 2 years
comparison of the percentages of correctly identified sound cues and the SNR corresponding to the subjective trade-off | 2 years
percentages of sound cues correctly identified by the participants using non-personalised speech enhancement strategies | 2 years
percentages of sound cues correctly identified by the participants using personalised speech enhancement strategies | 2 years
comparison of percentages of words correctly repeated | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CEntre de Recherche et d'Innovation en Audiologie Humaine, Paris, France

IPD SHARING:
Plan to Share IPD: No